CLINICAL TRIAL: NCT03590457
Title: The Impact of High-Flow Nasal Cannula on Swallow Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brady Scott, Associate Professor, Director of Clinical Education, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18012503
Record Dates: First submitted 2018-06-26; First posted 2018-07-18 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-08

CONDITIONS: Swallowing Disorder; Respiratory Insufficiency
MeSH Terms: conditions — Deglutition Disorders; Respiratory Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- High-Flow/Swallow (Other): All participants will be subjected to all three flows randomly. All participants will be asked swallow water and applesauce
  Interventions: Device: Airvo 2; High-Flow nasal cannula system

INTERVENTIONS:
Device: Airvo 2; High-Flow nasal cannula system — Noninvasive device used to deliver humidified oxygen at high flow rates up to 60 liters per minute

SUMMARY:
Background: High-flow nasal cannula (HFNC) is a non-invasive heated and humidified oxygen delivery device that is capable of delivering high-flow rates. It is a relatively new modality that has been introduced as an alternative to conventional oxygen therapy. The clinical value of the use of HFNC is not limited to its ventilation and oxygenation effects, it enables the patient to talk and is purported to permit oral feeding during oxygen therapy despite the limited evidence regarding its impact on swallow function. This study will determine the impact of different flow rates of a high-flow nasal cannula on spontaneous swallowing frequency at rest and swallowing effort and timing while swallowing. Methods: This is a prospective study designed to measure swallowing frequency and swallowing effort in fifty healthy adult volunteers. Participants will receive three levels of HFNC flow rates (30, 45, and 60 L/min) through nasal prongs. The study participants will be asked to swallow measured amounts of water and applesauce and subjected to each flow rate for 15 minutes. Swallowing effort measurement through surface electromyography (sEMG) will be recorded at baseline and the three levels of HFNC flow rates interventions.

DETAILED DESCRIPTION:
High-flow nasal cannula (HFNC) is a non-invasive heated and humidified oxygen delivery device that is capable of delivering up to 60 L/min of flow. It is a relatively new modality that has been introduced as an alternative to conventional oxygen therapy in patients with chronic obstructive pulmonary disease (COPD) respiratory failure, obstructive sleep apnea (OSA)6, post-extubation, and status asthmaticus The humidified gas preserves mucociliary function that prevents secretion retention and enhances patient's comfort. This feature allows prolonged use of HFNC in clinical sittings of up to 30 days

In addition to its ability to provide adequate humidification levels, HFNC has various respiratory physiological effects. These physiological effects include: alveolar recruitment, dead space washout, and decreased airway resistance. The clinical value of the use of HFNC is not limited to its ventilation and oxygenation effects, it enables the patient to talk and is purported to permit oral feeding during oxygen therapy.

Currently, despite the fact that patients are often permitted to eat while receiving HFNC therapy, there is insufficient evidence regarding the impact of HFNC on swallow function. The uncertainty of the effect of this oxygen delivery device on swallow function arises not only from the limited number of studies, but also the contradictory results. For example, Sanuki et al. reported that increasing the flow rates of the HFNC resulted in enhanced swallow function by reducing reflex latency. Based on their findings, the researchers suggested that the use of HFNC should not affect the decision to start or resume feeding. Similarly, Lader et al. proposed that the use of high-flow nasal cannula should not delay oral alimentation. On the contrary, Ferrara et al. conducted a study in neonates and concluded that providing feeding while using Nasal Continuous Positive Airway Pressure (nCPAP) increased the risk of aspiration. These opposing outcomes support the need for further studies to obtain more definitive evidence.

Methods:

Spontaneous Swallowing Frequency:

Spontaneous swallowing is an airway protection reflex and the measurement of its frequency is considered to be a sensitive indicator of swallow function. This index can sensitively identify dysphagia and other swallowing-related disorders. Furthermore, the reduction in this index is associated with increased level of secretions and chest infections. One modality used to measure swallowing frequency is surface electromyography (sEMG), which records electric activity during swallow via an electrode placed on the skin under the chin. This non-invasive technology has been used for more than 20 years to record various aspects of swallowing physiology. In this study, sEMG will be used because of its feasibility, accuracy, and ability to detect a swallow.

Swallowing Effort and Timing:

Swallowing effort via submental sEMG provides an objective measurement of lingual and sub-mental muscle activity during the act of swallowing. Measurements include muscle contraction amplitude and contraction timing/speed. Clinically, swallowing effort parameters have been used to document normative values in healthy individuals, as well as to document the effects of a disease on swallowing. Prior research has shown that both amplitude and timing are influenced by multiple factors including the volume and viscosity of the item (or bolus) being swallowed, and the age and gender of the person swallowing. However no study has investigated the effects of HFNC on either swallowing effort parameter.

The primary aim of this research is to determine the impact of different flow rates of a high-flow nasal cannula on spontaneous swallowing frequency at rest and swallowing effort and timing while swallowing.

This is a prospective study designed to measure swallowing frequency and swallowing effort in fifty healthy adult volunteers (25 participants will be between 21 and 49 years old; and the other 25 above 50 years old). To recruit volunteer participants, an email will be sent via university internal email system to the faculty, students and employees in the departments of Respiratory Care and Speech Language Pathology. Snowball sampling (non-probability sampling) will also be utilized to recruit individuals outside of those departments. No compensation is offered to the participants. Enrolled participants are sub-categorized into two different age groups to determine if there are any swallowing differences between the different age groups. Inclusion criteria include individuals who are older than 21 years of age and have no cognitive impairment. Exclusion criteria include individuals who are less than 21 years of age, have a history of dysphagia or disease/condition that may cause dysphagia, current use of medications that alter swallowing function, nasal obstruction, and the presence of a tracheostomy tube.

Upon meeting inclusion criteria, informed consent explaining the procedure and potential harm will be obtained and a copy will be given to the subject. Then, a unique identification code number will be assigned to protect the subject's identity.

HFNC:

The AIRVO 2 high-flow nasal cannula system (Fisher and Paykel Healthcare Limited, Panmure, Auckland, New Zealand) will be used. Nasal prongs sizes are chosen as per manufacturer recommendations. Participants will receive three levels of HFNC flow rates (30, 45, and 60 L/min) through nasal prongs. If a small-size nasal prong is used, the participant will receive 30, 45, and 50 L/min flow rates instead of 30, 45, and 60 L/min, as manufacturer recommendations state the maximum liter flow for a small-size nasal prong is 50 L/min. Oxygen concentration will be set at 21% and a temperature of 37 °C. First, individuals will be placed on the sEMG monitor. Following the application of the sEMG, each participant will sit quietly for 10 minutes, before being attached to the HFNC, so a baseline swallow frequency can be established. After the baseline swallow frequency is established, each participant will be asked to swallow 8 boluses: 2 trials of water at 2 volumes (5 and 10 mL) and 2 trials of applesauce at 2 volumes (5 and 10 mL). Participants will rest for 15 seconds after completing each swallow. This procedure will establish the participant's baseline swallowing effort measurements. Once these swallows have been completed, the participant will be placed on the HFNC. Each participant will be placed on three different flow rates (30, 45, and 60 L/min or 30, 45, and 50 L/min) in random order. The random order will be generated by an online random number tool (https://www.randomizer.org). The study participant will be subjected to each flow rate for 15 minutes. During the first 10 minutes, swallow frequency will be recorded. After 10 minutes at the given flow, the participant will complete the 8 aforementioned swallows. After completing all of the swallowing trials, the participant will be removed from the HFNC for a period of 10 minutes. This process will be repeated for all three flowrates for a total of 32 boluses swallowed.

Swallowing Frequency:

Swallowing frequency is analyzed by sEMG signals recorded on the KayPentax Digital Swallow Workstation™ with integrated digital swallowing signals lab (DSW™, Model 7120, New Jersey). A three-sensor sEMG electrode (Uni-Patch™, Disk #7500, Covidien Corporation, Tyco Healthcare, Wabasha, MN) will be placed on the anterior neck skin under the chin, over the submental muscles above the hyoid bone. Each patch will include two recording electrodes and a third ground electrode. Spontaneous swallowing frequency is calculated as the number of swallows per minute (SPM) for 10 minutes on room air and then for each HFNC intervention. Swallows will be counted from the visual myographic waveform produced by the DSW.

Swallowing Effort:

Both swallowing amplitude and timing parameters will be obtained by analyzing the individual graphic waveforms produced by the DSW algorithm. Measures will be obtained for each of the 8 swallows, at each of the HFNC flow rates.

Procedures Done for Research Purpose

The use of HFNC with three levels of flow (30, 45, and 60 L/min or 30, 45, and 50 L/min [for small-size nasal prongs]).

Swallow frequency measurement through sEMG.

Swallowing effort measurement through sEMG - participants will swallow measured amounts of water and applesauce. Presentation of the different volumes and viscosities will be done in pre-determined random order.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* No cognitive impairments

Exclusion Criteria:

* Less than 21 years old
* History of swallow dysphagia
* History of disease/condition that may cause dysphagia
* Use of medications that may alter swallow function
* Nasal obstruction
* Presence of tracheostomy tube

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Scott, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Flow/Swallow
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High-Flow/Swallow
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: data were not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Swallow Frequency Recorded by Surface Electromyography (sEMG)
Description: Number of swallows
Time Frame: each swallow frequency exam took 1 minute, exams were done for each flow rate which took up to 2 hours to complete
Population: swallow frequency
Measure: Mean (Standard Deviation); unit: number of swallows
Arm/Group | High-Flow/Swallow
Number analyzed (Participants) | 18
number of swallows
  swallow frequency at baseline | 1.12 (0.75)
  swallow frequency at 30 L/min | 1.13 (0.79)
  swallow frequency at 45 L/min | 3.91 (10.26)
  swallow frequency at 60 L/min | 1.01 (0.67)

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-Cause Mortality was not monitored/assessed
Arm/Group | High-Flow/Swallow
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03590457/Prot_SAP_000.pdf